CLINICAL TRIAL: NCT00178880
Title: MRI Imaging of Chronobiologic Abnormalities in Depression
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 010242
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Depression
Keywords: depression; MRI; imaging
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Healthy volunteers
- Depressed patients

SUMMARY:
The purpose of the study is to identify and understand patterns of brain activity when people are depressed. The study will use an imaging method called Magnetic Resonance Imaging (MRI) which does not involve any exposure to radioactivity or radioactive substances.

DETAILED DESCRIPTION:
The purpose of the study is to identify and understand patterns of brain activity when people are depressed. The study will use an imaging method called Magnetic Resonance Imaging (MRI) which does not involve any exposure to radioactivity or radioactive substances.

ELIGIBILITY:
Inclusion Criteria:

* WEIGHT: less than or at 20% over ideal weight, as specified in the 1983 Metropolitan Height and Weight Tables. Patients who deviate from these ranges may be reviewed on an individual basis by the Investigator. This criterion is necessary because of mechanical limitations in fitting overweight individuals into the scanner, and the risk of excessive claustrophobic responses if tightly constricted.
* HEALTH: healthy, ambulatory normal or depressed adults

Exclusion Criteria:

* Presence of aneurysm clips, cardiac pacemakers, cochlear implants, metal in the eyes, and implanted insulin pumps.
* Evidence of significant hepatic, gastrointestinal, renal, respiratory, endocrine, hematologic, neurologic, psychiatric, or cardiovascular system abnormalities.
* Pregnancy.
* Patients with a known or suspected history of alcohol or drug misuse and/or a positive urine drug screen.
* Patients who are unwilling or unable to abide by the requirements of the study or who violate the prohibitions and restrictions of the study.
* Any condition which would make the patient, in the opinion of the Investigator, unsuitable for the study.
* Patients on antidepressants may not be taking any other medication, except at the discretion of the investigator. Untreated depressed or healthy subjects must be free of all medications except as approved by the investigator.
* Patients with serious medical illness, history or signs/symptoms of lumbar spine/disc disease or significant laboratory findings.
* Patients who present significant suicide risk, e.g. with a history of highly impulsive suicide attempts.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers and depressed patients.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2008-11 (Actual); Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Salomon, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States